CLINICAL TRIAL: NCT06387784
Title: Acute Effect of Beetroot Juice Supplementation in Pregnant Women With Pre-eclampsia: a Single-Blind Randomized Placebo-Controlled Trial
Brief Title: Acute Beetroot Juice Supplementation in Pre-eclampsia Pregnancies
Acronym: BEET_PE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Hospital das Clínicas de Ribeirão Preto (Other); Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Ricardo de Carvalho Cavalli, Professor Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/823
Record Dates: First submitted 2024-04-16; First posted 2024-04-29 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Pre-Eclampsia
Keywords: Pre-eclampsia; Pregnancy; Beetroot Juice; Nitric Oxide
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, single-blind, parallel-group study assessing acute rich-nitrate juice on pregnant women diagnosed with early and late-onset pre-eclampsia. Participants will be divided into four distinct groups: two groups for each onset category. Within each group, participants will be further divided into a control group and a treated group. The assignment of participants to these groups will be randomized using an online program.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Early-onset pre-eclampsia beetroot juice (Experimental): A single dose of 70 ml of nitrate-rich beetroot juice containing 400 mg of nitrate.
  Interventions: Dietary Supplement: Beetroot juice
- Early-onset pre-eclampsia placebo juice (Placebo Comparator): A single dose of 70 ml of a formulation with a similar taste, smell, and texture.
  Interventions: Dietary Supplement: Placebo juice
- Late-onset pre-eclampsia beetroot juice (Experimental): A single dose of 70 ml of nitrate-rich beetroot juice containing 400 mg of nitrate.
  Interventions: Dietary Supplement: Beetroot juice
- Late-onset pre-eclampsia placebo juice (Placebo Comparator): A single dose of 70 ml of a formulation with a similar taste, smell, and texture.
  Interventions: Dietary Supplement: Placebo juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — In the morning, pregnant women with pre-eclampsia will consume a single dose of 70 ml of nitrate-rich beetroot juice containing 400 mg of nitrate. Participants will be monitored to assess the acute effects of nitrate intake for 6 hours.
  Arms: Early-onset pre-eclampsia beetroot juice; Late-onset pre-eclampsia beetroot juice
Dietary Supplement: Placebo juice — In the morning, pregnant women with pre-eclampsia will consume 70 ml of a placebo juice. The placebo juice will be similar in appearance and taste to the nitrate-rich beetroot juice. Participants will be monitored to compare the acute effects of beetroot juice with the placebo intake for 6 hours.
  Arms: Early-onset pre-eclampsia placebo juice; Late-onset pre-eclampsia placebo juice

SUMMARY:
Pre-eclampsia is a serious condition that typically affects pregnant women after the 20th week of pregnancy, characterized by high blood pressure and damage to organs such as the kidneys and liver. Currently, treatment options are limited, which has prompted researchers to explore alternative approaches. One such promising alternative is dietary nitrate found in vegetables like beetroot, as nitrate can be converted into nitric oxide in the body, which helps lower blood pressure. This study aims to determine the acute effects of nitrate-rich beetroot juice on blood pressure, several blood and salivary markers in pregnant women with pre-eclampsia. Furthermore, the study will assess fetal blood flow using Doppler ultrasound. The investigators want to understand the kinetics of nitrate and nitric oxide metabolites and assess the temporal dependency of the hypotensive response. Through this investigation, the investigators seek evidence of nitrate-enriched beetroot juice as an adjunct therapy in managing pre-eclampsia.

DETAILED DESCRIPTION:
The study will include women diagnosed with either early-onset pre-eclampsia or late-onset pre-eclampsia, following the guidelines of the American College of Obstetricians and Gynecologists. Participants will be required to sign informed consent forms following a thorough explanation of the study. A total of four groups will be established, with twenty-four pregnant women randomly assigned to each group using a free online program. In each group (early-onset and late-onset pre-eclampsia), forty-eight pregnant women will receive nitrate-enriched beetroot juice (Beet It®, James White, UK), while another forty-eight will receive an equivalent amount of placebo juice. The trial will commence in the morning, between 7:30 and 8:30 am, after a standardized, low-nitrate breakfast provided by the hospital. Participants will be instructed to avoid nitrate-rich foods the previous evening and will receive guidance from the project team and the hospital's nutrition service. The hospital's nutritional team will oversee the dietary procedures. Ambulatory blood pressure monitoring will be conducted for six hours following the ingestion of juice or placebo. Saliva samples will be collected to assess nitrate reductase activity, and blood samples will be drawn to measure nitrate, nitrite, and nitrosothiol (nitric oxide metabolites), as well as to perform biochemical analyses of oxidative stress. Doppler ultrasound and Doppler velocimetry evaluation will be conducted at the peak action time of nitrate, which is estimated to occur two hours post-ingestion, based on previous research.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at or beyond the 20th week of gestation.
* Hospitalized at Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto.
* Diagnosed with early or late-onset pre-eclampsia confirmed by a medical professional.
* Capacity to provide written informed consent for study participation.

Exclusion Criteria:

* Multiple pregnancies.
* Uncontrolled arterial hypertension (Systolic Blood Pressure > 160 mmHg or Diastolic Blood Pressure > 100 mmHg).
* Pregnant women with a body mass index > 40 kg/m²
* Severe gestational complications.
* History of food allergy with hypersensitivity to beetroot.
* Smokers.
* Chronic alcohol consumption.
* Use of medications, except for antihypertensive.
* Diagnosis of renal or hepatic disease affecting nitrate metabolism.
* Cardiac conditions such as moderate to severe congestive heart failure and coronary artery disease.
* Pre-existing type 1 or type 2 diabetes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Acute Effect of Beetroot Juice Supplementation on Blood Pressure | Every 30 minutes up to 6 hours post-supplementation.
  Assessment of the acute effect of beetroot juice supplementation on blood pressure (measured in millimetres of mercury - mmHg) in pregnant women diagnosed with early and late-onset pre-eclampsia, measured every 30 minutes up to 6 hours post-supplementation, starting 30 minutes before ingestion, compared to a placebo group.

SECONDARY OUTCOMES:
Plasma Concentrations of Nitric Oxide Metabolites | At baseline and up to 6 hours post-supplementation.
  Assessment of plasma concentrations of nitric oxide metabolites (nitrite, nitrate and nitrosothiol) in pregnant women diagnosed with pre-eclampsia, comparing those receiving beetroot juice supplementation and those receiving placebo.
Concentration of Salivary Nitrate Reductase Enzyme | At baseline and up to 6 hours post-supplementation.
  Assessment of the activity of the nitrate reductase enzyme in saliva in each study group.
Plasma Lipid Peroxidation Levels | At baseline and up to 6 hours post-supplementation.
  Assessment of the degree of lipid peroxidation, measured by the level of malondialdehyde in each study group.
Concentration of Total Antioxidant Capacity in Plasma | At baseline and up to 6 hours post-supplementation.
  Determination of the plasma concentration of total antioxidant capacity of plasma, measured in Trolox equivalent antioxidant capacity, in each study group.
Maternal Blood Flow Velocity | 2 hours post-supplementation of beetroot juice or placebo.
  Maternal blood flow velocity will be measured in centimeters per second (cm/s) using Doppler ultrasound, in each study group.
Fetal Heart Rate | 2 hours post-supplementation of beetroot juice or placebo.
  Fetal heart rate will be measured in beats per minute (bpm) using Doppler ultrasound, in each study group.
Umbilical Arterial Pulsatility Index | 2 hours post-supplementation of beetroot juice or placebo.
  The umbilical arterial pulsatility index will be calculated and reported as a percentile, in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo C Cavalli, Dr, Principal Investigator — Medical School of Ribeirao Preto, USP
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
We will provide access to individual de-identified participant data and related study documents upon request from qualified researchers, subject to certain criteria, conditions, and exceptions.